CLINICAL TRIAL: NCT03694015
Title: SUPR-3D: A Randomized Phase III Trial Comparing Simple Unplanned Palliative Radiotherapy Versus 3D Conformal Radiotherapy for Patients With Bone Metastases
Brief Title: SUPR-3D: Simple Unplanned Palliative Radiotherapy Versus 3D Conformal Radiotherapy for Patients With Bone Metastases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Robert Olson, Radiation Oncologist & Department Head Radiation Oncology & Developmental Radiotherapeutics, British Columbia Cancer Agency
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUPR-3D
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Neoplasm Metastasis; Neoplastic Processes; Neoplasms; Pathologic Processes
MeSH Terms: conditions — Neoplasm Metastasis; Neoplastic Processes; Neoplasms; Pathologic Processes

STUDY DESIGN:
Intervention Model Description: Simple randomization with stratification will be used to randomly assign patients to either Arm 1 or Arm 2 in a 1:1 ratio using a computer-generated randomization scheme.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SUPR (Arm 1) (Active Comparator): Planning according to local protocols. No more than 2 fields; no beam modifying devices, other than multileaf collimators (MLCs). Alternate weighting of beams allowed (ie. 1:2 AP:PA). Review of dosimetry not required, if performed as per institutional standard.
  Minimum of kV image matching on unit daily.
  Interventions: Radiation: SUPR
- VMAT rapid (Arm 2) (Active Comparator): Contouring: GTV based on available imaging (CT sim scan alone-no special imaging), expect to be between 1.5cm and 20cm clinically or from imaging. CTV-optional in all scenarios. If using CTV=GTV +0.5 to 0.7cm adjust to anatomy as follows:
  * If only bone involved: recommend not to expand past bone; but a 0.5-0.7cm CTV expansion outside of bone into muscle or soft tissue is allowed at RO discretion
  * If bone and soft tissue involved: 0.5 to 0.7cm CTV expansion is optional, allowed at RO discretion
  * If spinal metastases: CTV is optional. If used can include whole vertebral body at RO discretion PTV=CTV or GTV+(1 to 1.5)cm at RO discretion. PTV_eval=PTV cropped 0.5cm below skin. OARs: max 2 OARs permitted for VMAT arm. OAR constraints are at RO discretion. If lung/kidneys are within 5cm of PTV, absence of constraints for contours should be noted in treatment plans or dose constraint sheet prior to planning. PTV can be compromised for OAR at RO's discretion. Kidneys considered 1 organ
  Interventions: Radiation: VMAT

INTERVENTIONS:
Radiation: SUPR — simple unplanned palliative radiotherapy-(either 8 Gy in 1 fraction or 20 Gy in 5 fractions), chosen pre-randomization at ROs or centres discretion
  Arms: SUPR (Arm 1)
Radiation: VMAT — volumetric modulated arc therapy--(either 8 Gy in 1 fraction or 20 Gy in 5 fractions), chosen pre-randomization at ROs or centres discretion
  Arms: VMAT rapid (Arm 2)

SUMMARY:
The primary objective is to patient-reported Quality of Life related to complete control of Radiation Induced Nausea and Vomiting (RINV) between standard palliative radiotherapy and VMAT. Secondarily, we will assess rate of complete control of RINV. However, the investigators hypothesize that there will be no difference in pain response between the two arms, because they are receiving the same dose.

DETAILED DESCRIPTION:
For this study, SUPR (simple unplanned palliative radiotherapy) refers to the delivery of radiation to the treatment area with a simple technique, either two opposed fields (parallel opposed pair), or a single direct field. The entire portal is exposed to the specified dose and therefore does not spare normal tissue. This technique requires minimal calculation, and typically the dose distribution is not reviewed by the radiation oncologist or medical physics.

In general, the adverse event profile of RT is associated with irradiation of normal tissue within the treatment field. With the dose prescribed in this study, the probability of serious adverse effects is exceedingly low. However, fatigue, soreness, pain flare, and skin-redness in the irradiated area are relatively common adverse events. In addition, site-specific toxicity could occur, including esophagitis, nausea, or diarrhea when there is dose delivered to the GI tract. Avoiding this toxicity is a motivating factor for the study.

In order to deliver 3D Conformal Radiotherapy, a computerized tomography (CT) simulation is used to develop the treatment plan. The goal is to deliver a conformal radiation dose to the target volume with maximal sparing of the normal tissue. VMAT (Volumetric Modulated Arc Therapy) is a type of 3D conformal RT, and delivers the radiation dose more conformally than SUPR, possibly reducing acute and late toxicity. The disadvantages of VMAT include more complex planning and quality assurance processes compared with SUPR. The complex planning required can be time-consuming, which can have a significant impact on departmental resources, and the wait time for the patient.

Bone metastases are the most common site of distant metastases and can cause severe and disabling effects, including pain, spinal cord compression and pathologic fracture. These complications can greatly affect a patient's quality of life and cause immense suffering.

Radiotherapy (RT) is an effective treatment for palliative patients with painful bone metastases. It is also efficacious in preserving function and maintaining skeletal integrity, while minimizing the occurrence of adverse skeletal related events. There is a significant amount of evidence showing that a single fraction (SF) of RT provides equivalent pain relief as multiple fractions (MF), which are associated with more acute toxicity, are less convenient for patients and costlier for the health care system. Therefore, single fraction radiation therapy (SFRT) is encouraged, but 20 Gy in 5 fractions is also allowed in this study, though should be chosen only in patients with a complicated bone metastases by fracture, neurological deficit (e.g. spinal cord compression), or a large soft tissue component. In patients with advanced disease, management strategies focus on improving quality of life (QOL), rather than conventional endpoints such as survival.

Currently, the standard of care in British Columbia for palliative patients with bone metastases is SUPR. In other jurisdictions, however, factors such as physician remuneration make other complex planning techniques more popular.

BC Cancer is publicly funded with no direct costs to patients. All RT in the province is provided by 6 centres where radiation oncologists receive an annual salary, which are independent of RT treatment technique and duration. Due to the lack of financial incentive associated with a more complex RT plan, BC Cancer is a unique clinical setting to assess the use of VMAT versus SUPR.

As facilities providing RT have gained more experience with VMAT and improvements to VMAT planning software have been made, the planning time required has been reduced. Previously, approximately 2 weeks was required for a team at the BC Cancer to create a VMAT plan for a palliative patient with bone metastases; however, we hypothesize this can now be reduced to three days in settings with low dose prescription.

This study will allow the investigators to determine if there is reduced toxicity associated with VMAT compared to SUPR with only a modest impact on resources. The investigators hypothesis is that VMAT will have reduced toxicity compared with SUPR for palliative patients with bone metastases. The investigators also hypothesize that there will be no difference between the two arms in terms of pain response, due to the fact that the doses are equal. This hypothesis is driven by the radiobiologic rationale, which defines effective RT as the ability of radiation to induce tumour cell death while sparing normal cells.

The importance in determining if there is any benefit in terms of toxicity with VMAT compared with SUPR for palliative patients with bone metastases is obvious when consequences related to its adoption are considered. As previously discussed, although the planning time has been drastically reduced, there is still an expected modest increase in resources required to carry out a VMAT plan. For patients, the pre-treatment process of VMAT is more burdensome, i.e. patients have to wait longer before receiving VMAT as compared to SUPR, due to the increased plan complexity. Therefore, it is important to consider the patient experience in relation to the RT administration.

In summary, evidence that either supports or refutes the hypothesis that VMAT will have reduced toxicity compared with SUPR for patients with bone metastases will be helpful in guiding future practices. We are not aware of any other randomized control trials (completed or ongoing) that have addressed this issue, though a London Ontario study is randomizing patients receiving palliative lung RT to SUPR vs VMAT. Due to the implications of VMAT on departmental resources and patient experience, better evidence from a randomized control trial is required before the widespread use of this technique can be justified.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Able to provide informed consent
* Clinical diagnosis of cancer with bone metastases (biopsy not required)
* Currently being managed with palliative intent RT to 1-3 RT fields for bone metastases, at least one RT field (PTV) must (at least) partly lie within T11-L5 or pelvis.
* ECOG Performance Status 0-3
* Patient has been determined to potentially benefit from 8 Gy or 20 Gy
* Radiation Oncologist is comfortable prescribing 8 Gy in 1 fraction or 20 Gy in 5 fractions RT for bone metastases
* Negative pregnancy test result for women of child-bearing potential
* The baseline assessment must be completed within required timelines, prior to randomization.
* Patients must be accessible for treatment and follow-up. Investigators must assure themselves the patients randomized on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.
* For simplicity of planning, expected GTV should be less than 20 cm based on radiological or clinical evidence
* Patient must be prescribed a 5-HT3 receptor antagonist (e.g. Ondansetron) as antiemetic prophylaxis prior to RT start.
* Patient is able and willing to complete the quality of life questionnaires, and other assessments that are a part of this study, via paper or using PatientPortals.ca or REDCap if they provide their email address on the informed consent

Exclusion Criteria:

* Serious medical co-morbidities precluding radiotherapy
* Clinical evidence of spinal cord compression
* Spinal cord in treatment field has already received at least >30 Gy EQD2
* Whole brain radiotherapy (WBRT) within 4 weeks of RT start or planned WBRT in the first 4 weeks after last RT
* Solitary plasmacytoma
* Pregnant or lactating women
* Target volume cannot be encompassed by a single VMAT isocentre
* Custom mould room requirements (shells and other immobilization that is standard-of-care is acceptable)
* Greater than two organs-at-risk requiring optimization.
* Patients requiring treatments outside standard clinical hours
* Implanted electronic device within 10 cm of the RT fields
* Prostheses in the axial plane of the target, or within 1 cm of the PTV out-of-plane
* Previous RT that requires an analysis of cumulative dose (i.e. sum plans or EQD2 calculations)
* Oral or IV contrast if the local standard-of-care requires compensation for this in planning.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-12-02 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Reported Quality of life related to Radiation Induced Nausea and Vomiting (RINV) | day 1-5
  RINV as measured by the Functional Living Index - Emesis (FLIE) at day 5 post RT start

SECONDARY OUTCOMES:
Control of RINV Radiation Induced Nausea and Vomiting (RINV) | day 1-5
  as measured by a daily patient diary (day 1-5)
Patient Reported Pain Response | baseline, 2 weeks, and 4 weeks post treatment
  as measured by the Brief Pain Inventory
Patient Reported Use of Medications | baseline, 2 weeks, and 4 weeks post treatment
  as measured by the Patient Diary
Patient Reported Fatigue, Nausea, Vomiting | baseline, 2 weeks, and 4 weeks post treatment
  as measured by the PRO-CTCAE
Patient Reported Quality of Life | baseline, 2 weeks, and 4 weeks post treatment
  as measured by EORTC QLQ C-15 PAL
Economic Analysis | baseline, 2 weeks, and 4 weeks post treatment
  as measured by EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Rob Olson, MD, Principal Investigator — British Columbia Cancer Agency
Locations (5):
- Canada (5):
  - BC Cancer, Prince George, British Columbia
  - BC Cancer, Vancouver, British Columbia
  - BC Cancer - Victoria, Victoria, British Columbia
  - London Health Sciences Centre, London, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teoh M, Clark CH, Wood K, Whitaker S, Nisbet A. Volumetric modulated arc therapy: a review of current literature and clinical use in practice. Br J Radiol. 2011 Nov;84(1007):967-96. doi: 10.1259/bjr/22373346. PMID 22011829
- [Background] Webb S. Advances in treatment with intensity-modulated conformal radiotherapy. Tumori. 1998 Mar-Apr;84(2):112-26. doi: 10.1177/030089169808400206. PMID 9620234
- [Background] Guerrero Urbano MT, Nutting CM. Clinical use of intensity-modulated radiotherapy: part I. Br J Radiol. 2004 Feb;77(914):88-96. doi: 10.1259/bjr/84246820. PMID 15010378
- [Background] Miles EA, Clark CH, Urbano MT, Bidmead M, Dearnaley DP, Harrington KJ, A'Hern R, Nutting CM. The impact of introducing intensity modulated radiotherapy into routine clinical practice. Radiother Oncol. 2005 Dec;77(3):241-6. doi: 10.1016/j.radonc.2005.10.011. Epub 2005 Nov 17. PMID 16298002
- [Background] Chow E, Zeng L, Salvo N, Dennis K, Tsao M, Lutz S. Update on the systematic review of palliative radiotherapy trials for bone metastases. Clin Oncol (R Coll Radiol). 2012 Mar;24(2):112-24. doi: 10.1016/j.clon.2011.11.004. Epub 2011 Nov 29. PMID 22130630
- [Background] Lutz S, Berk L, Chang E, Chow E, Hahn C, Hoskin P, Howell D, Konski A, Kachnic L, Lo S, Sahgal A, Silverman L, von Gunten C, Mendel E, Vassil A, Bruner DW, Hartsell W; American Society for Radiation Oncology (ASTRO). Palliative radiotherapy for bone metastases: an ASTRO evidence-based guideline. Int J Radiat Oncol Biol Phys. 2011 Mar 15;79(4):965-76. doi: 10.1016/j.ijrobp.2010.11.026. Epub 2011 Jan 27. PMID 21277118
- [Background] Nielsen OS. Palliative radiotherapy of bone metastases: there is now evidence for the use of single fractions. Radiother Oncol. 1999 Aug;52(2):95-6. doi: 10.1016/s0167-8140(99)00109-7. No abstract available. PMID 10577693
- [Derived] Olson R, Schlijper R, Chng N, Matthews Q, Arimare M, Mathews L, Hsu F, Berrang T, Louie A, Mou B, Valev B, Laba J, Palma D, Schellenberg D, Lefresne S. SUPR-3D: A randomized phase iii trial comparing simple unplanned palliative radiotherapy versus 3d conformal radiotherapy for patients with bone metastases: study protocol. BMC Cancer. 2019 Oct 28;19(1):1011. doi: 10.1186/s12885-019-6259-z. PMID 31660894

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/15/NCT03694015/Prot_SAP_005.pdf